CLINICAL TRIAL: NCT05224544
Title: Exploratory Study Investigating the Acute Effect of Intermittent Catheterization on the Bladder Mucosa of Healthy Volunteers With a Prototype Micro Hole Zone Catheter Compared to a Conventional 2-eyelet Catheter
Brief Title: Intermittent Catheterisation on the Bladder Mucosa of Healthy Volunteers With a Prototype Micro Hole Zone Catheter
Acronym: CP341
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CP341
Record Dates: First submitted 2021-12-03; First posted 2022-02-04 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Prototype Catheter (Experimental): Healthy volunteers to test the prototype intermittent catheter with a microhole zone.
  Interventions: Device: Investigational prototype device
- Comparator Catheter (Active Comparator): Healthy volunteers to test the comparator intermittent catheter with two conventional eyelets.
  Interventions: Device: Comparator device

INTERVENTIONS:
Device: Investigational prototype device — The test product is a urinary catheter for bladder drainage through the urethra. The product is for intermittent use.
  Other Names: prototype microhole zone catheter
  Arms: Prototype Catheter
Device: Comparator device — The comparator is a urinary catheter for bladder drainage through the urethra.
  Other Names: "Infyna chic"
  Arms: Comparator Catheter

SUMMARY:
This investigation is a randomized, single-blinded, parallel, single-center investigation. In total, up to 50 subjects (40 completers) were included and each subject had two test visits overseen by the Principal Investigator (PI), or designee. Each subject were enrolled in the investigation, which lasted up to 3 days (if Day 0 and Day 1 were not on same day). The subjects were randomly assigned to test either the prototype product or the comparator product, with at least 20 subjects assigned to each product.

DETAILED DESCRIPTION:
This investigation was a randomized, single-blinded, parallel, single-center investigation. Up to 50 subjects (40 completers) will be included and each subject will have two test visits overseen by the Principal Investigator (PI), or designee. Each subject will be enrolled in the investigation, which can be up to 3 days (if Day 0 and Day 1 are not on same day). The subjects will be randomly assigned to test either the prototype product or the comparator product, with at least 20 subjects assigned to each product. The subjects will undergo cystoscopy and catheterization.

ELIGIBILITY:
Inclusion Criteria:

1. Has given written informed consent
2. Is at least 18 years and have full legal capacity
3. Is female
4. Has a negative urine Multistix dipstick test for erythrocytes (haematuria)

Exclusion Criteria:

1. Has used an internal urinary catheter or cystoscopy within the past month
2. Has prior history of bladder surgery
3. Is symptomatic and/or on medication for overactive bladder
4. Has evidence of ongoing, active, symptomatic urinary tract infection (UTI) (assessed by PI, or delegate)
5. Is pregnant and/or breast-feeding
6. Is participating in other clinical investigations during this investigation
7. Is menstruating during study period

Ages: 18 Years to 110 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This device is a female catheter.
Enrollment: 43 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Selwyn Spangenthal, MD, Principal Investigator — American Health Research
Locations (1):
- American Health Research, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Prototype Catheter: Healthy volunteers to test the prototype intermittent catheter.
  Prototype device: The test device is a urinary catheter for bladder drainage through the urethra. The product is for intermittent use.
- Comparator Catheter: Healthy volunteers to test the comparator.
  Comparator: The comparator is a urinary catheter for bladder drainage through the urethra for intermittent use.
Period: V1, Visualization of the Bladder
Arm/Group | Prototype Catheter | Comparator Catheter
Started | 21 | 22
Completed | 21 | 22
Not Completed | 0 | 0
Period: V2, Catheterization and Visualization
Arm/Group | Prototype Catheter | Comparator Catheter
Started | 21 | 22
Completed | 19 | 21
Not Completed | 2 | 1
Not completed — Adverse Event | 2 | 1

BASELINE CHARACTERISTICS:
Population: Female healthy volunteers with an average age of 40 (range: 18-71 years) and no prior prophylactic antibiotic.
Groups:
- Prototype Catheter: Healthy volunteers to test the prototype investigational intermittent catheter.
  Test Catheter: The test product is a urinary catheter for bladder drainage through the urethra. The product is for intermittent use.
- Comparator Catheter: Healthy volunteers to test the comparator catheter.
  Comparator catheter: The comparator is a urinary catheter for bladder drainage through the urethra, for intermittent use.
- Total: Total of all reporting groups
Arm/Group | Prototype Catheter | Comparator Catheter | Total
Number analyzed (Participants) | 21 | 22 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (14.7) | 38.4 (16.7) | 39.7 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 43
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Prophylactic antibiotics [Count of Participants; unit: Participants] | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Appearance of the Bladder Mucosa (∆=Pre-catheterisation at Baseline and Post-catheterization and Visit 2) Rated on a 4-point Scale.
Description: Change in appearance of the bladder mucosa (∆=pre-catheterisation at baseline and post-catheterization and visit 2) rated on a 4-point scale.
  The 4-point scale defined as such:
  1. no lesions evident;
  2. minor mucosal and blood vessel lesions;
  3. major blood vessel lesions, and
  4. major mucosal and blood vessel lesions,
Time Frame: 2 days
Population: Intention to treat (ITT)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Change in Bladder Mucosa Pre- and Post-catheterization for the Prototype Catheter: Change in appearance of the bladder mucosa with prototype catheter, post- and pre-catheterization (∆), rated on a 4-point scale of:
  1. no lesions evident;
  2. minor mucosal and blood vessel lesions;
  3. major blood vessel lesions, and
  4. major mucosal and blood vessel lesions, post-catheterization (Visit 2).
- Change in Bladder Mucosa Pre- and Post-catheterization for the Comparator Catheter: Change in appearance of the bladder mucosa with comparator catheter, post- and pre-catheterization (∆), rated on a 4-point scale of:
  1. no lesions evident;
  2. minor mucosal and blood vessel lesions;
  3. major blood vessel lesions, and
  4. major mucosal and blood vessel lesions, post-catheterization (Visit 2).
Arm/Group | Change in Bladder Mucosa Pre- and Post-catheterization for the Prototype Catheter | Change in Bladder Mucosa Pre- and Post-catheterization for the Comparator Catheter
Number analyzed (Participants) | 19 | 21
score on a scale | 0.84 [0.58 to 1.11] | 0.76 [0.51 to 1.01]

ADVERSE EVENTS:
Time Frame: The study consisted of one inclusion visit (Visit 0) and two test visits (Visits 1 and 2) of approximately 1-2 hrs. The inclusion visit, and the first test visit were completed on the same day, when possible, and in those circumstances took two days to complete. For participants where V0 and V1 were not performed on the same days, the study took three days.
Groups:
- Prototype Catheter: Adverse event upon catheterization with prototype catheter
- Comparator Catheter: Adverse event upon catheterization with comparator catheter
Arm/Group | Prototype Catheter | Comparator Catheter
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21
Other Adverse Events (participants affected / at risk) | 9/19 | 2/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prototype Catheter (N=19) | Comparator Catheter (N=21)
Hematuria (Renal and urinary disorders) | 7 (7) | 1 (1) — Hematuria either pre- or post-catheterization
Urinary tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Burning sensation (Renal and urinary disorders) | 1 (1) | 0 (0) — Burning sensation during normal micturition
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Nausea due to antibiotic

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/44/NCT05224544/Prot_SAP_002.pdf